CLINICAL TRIAL: NCT07219927
Title: Real-World Patient Experiences Using Continuous Subcutaneous Apomorphine Infusion (ONAPGOTM) in the United States: A Prospective, Phase 4, Multicenter, Observational Study in Parkinson's Disease
Brief Title: Real-World Patient Experiences Using Continuous Subcutaneous Apomorphine Infusion (ONAPGOTM) in the United States:
Status: Recruiting | Type: Observational
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 830P401
Record Dates: First submitted 2025-06-09; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: ONAPGO
MeSH Terms: conditions — Parkinson Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Continuous Subcutaneous Apomorphine Infusion (ONAPGOTM)

SUMMARY:
Real-World Participants Experiences Using Continuous Subcutaneous Apomorphine Infusion (ONAPGOTM) in the United States: A Prospective, Phase 4, Multicenter, Observational Study in Parkinson's Disease

DETAILED DESCRIPTION:
This observational study includes an Enrollment Day (participants enrolled any time between their prescription for the infusion and ONAPGO initiation); a Baseline Period (prior to ONAPGO initiation which includes in-home education on the use of ONAPGO by the Clinical Nurse Navigator [CNN] according to standard practice for patients with PD-prescribed ONAPGO); Dose Initiation, Titration, and Optimization per Prescription Periods; a Maintenance Period; Maintenance CNN standard of care visits; and an End-of-Study (EOS)/Discontinuation Visit.

ELIGIBILITY:
Inclusion Criteria:

Participant has received a prescription for ONAPGO™ according to the standard of care.

Participant has opted into receiving support services from the Clinical Nurse Navigator (CNN), a registered nurse specially trained to work with persons with Parkinson's disease, as noted on the Prescription Enrollment Form.

The HCP/Investigator determines the participant is an appropriate study participant.

Participant is able and willing to provide informed consent (or informed assent form [IAF], as applicable) and signs the consent form on the Enrollment Day.

Exclusion Criteria:

Did not receive a prescription for ONAPGO™.

Prescribed ONAPGO™, but the HCP/Investigator determines the participant should not participate in this observational study.

Concomitant use of ONAPGO™ with 5-HT3 antagonists, including antiemetics (e.g., ondansetron, granisetron, dolasetron, palonosetron) or alosetron.

Known hypersensitivity to apomorphine or to excipients of ONAPGO™, including sulfite (e.g., sodium metabisulfite).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are eligible for participation in this study after they have received a prescription for Onapgo
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Titration Duration and Time to Optimized Dose | Approximately 52-60 weeks
  The time from the date of ONAPGO™ initiation to the date of Dose Optimization Confirmation, as documented by the HCP/Investigator Unit of Measure: days
Concomitant Parkinson's Disease (PD) Medication Adjustments | Approximately 52-60 week
  Percentage of participants requiring ≥1 adjustment to their concomitant PD medications, as documented by the HCP/Investigator. "Percentage of participants"
The number of titration visits or dose adjustments required to reach the final optimized dose. This is a count of a specific event | Approximately 52-60 weeks
  Number of titration visits or infusion adjustments to reach final optimized dose; Unit of Measure: count per participant

SECONDARY OUTCOMES:
Perception of Patient Global Health Improvement | Approximately 52-60 weeks
  Change from baseline in the Patient Global Impression of Change (PGI-C) scale, with scores ranging from 1 ("very much improved") to 7 ("very much worse"); lower scores indicate better outcomes. Unit of Measure: PGI-C score (range 1-7)
Caregiver Burden | Approximately 52-60 weeks
  Change from baseline in caregiver quality of life (QoL) as determined by scores on the European Quality of Life 5 Dimensions (EQ-5D) scale. This scale measures health-related QoL, with scores ranging from 0 (death) to 1 (full health). A higher score indicates a better outcome.
HCP/Investigator burden for ONAPGO providers | Approximately 52-60 weeks
  Change from baseline to each time point in scores over time on the modified 8-item HCP Burden Scale to assess the HCP perceived burden of managing patients on ONAPGO treatment
Evaluation of ONAPGO usage during the maintenance period | Approximately 52-60 weeks
  Hourly modal infusion rate (mg/hour) during the maintenance period Daily modal dose (mg/day) during the maintenance period Daily modal duration (hour) during the maintenance period
Safety by monitoring adverse events (AEs) | Approximately 52-60 weeks
  Safety is measured by AE evaluation according to the standard of care and the percentage of participants who discontinue ONAPGO™ treatment due to AEs

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Grall, PhD ANP-BC, Study Chair — Supernus Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Parkinson's Disease and Movement Disorders Center - Orange County (South), Aliso Viejo, California
  - Parkinson's Disease and Movement Disorders Center - Orange County (North), Irvine, California
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - Parkinson's Disease & Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Parkinson's Disease and Movement Disorders Center - Long Island, Commack, New York

IPD SHARING:
Plan to Share IPD: No